CLINICAL TRIAL: NCT01525758
Title: Eight-week, Multi-centre, Dose-response, Double Blind, Placebo-controlled, Randomized, Parallel-group, PhaseⅡ Trial to Evaluate Efficacy and Safety of SI000413 in Patients With Knee Osteoarthritis
Brief Title: Study of SI000413 in Knee Osteoarthritis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI000413_OA_Ⅱ
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — SI 000413; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SI000413 400mg (Experimental): tablet, SI000413 200mg bid
  Interventions: Drug: SI000413
- SI000413 600mg (Experimental): tablet, SI000413 200mg tid
  Interventions: Drug: SI000413
- SI000413 800mg (Experimental): SI000413 200mg, 2T bid
  Interventions: Drug: SI000413
- placebo (Placebo Comparator): placebo 2T tid for 8 weeks
  Interventions: Drug: microcrystalline cellulose

INTERVENTIONS:
Drug: SI000413 — 1 Tablet = 200mg, (400mg, 600mg or 800mg vs. placebo) for 8weeks
  Arms: SI000413 400mg; SI000413 600mg; SI000413 800mg
Drug: microcrystalline cellulose — identical number of tablets to active drug groups
  Other Names: SI000413 placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of SI000413 in patients with knee osteoarthritis by orally administration and to determine optimal dose.

DETAILED DESCRIPTION:
This is a dose-response, double blind , placebo-controlled study. All patients are required to have 2 weeks washout period from prior medication. Subjects will discontinue current medications 2 weeks prior to randomization. Among those who meet the inclusion criteria, only subjects recording visual analogue scale(VAS) of higher than 40mm(VAS range from 0mm(no pain) to 100mm(unbearable pain)) are enrolled in this study.

Subjects meeting screening criteria will be randomized to receive 8 weeks dosing of an active dose of SI000413 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 35-75 years old
2. Subjects must have a clinical or radiographic diagnosis of primary OA of the knee (diagnosed according to the ACR)

   * The presence of knee pain
   * At least one of the following

     * age older than 50 years
     * morning stiffness lasting less than 30 minutes
     * crepitus with motion
3. Subjects must have been symptomatic for at least 3 months prior to enrollment.
4. Subjects must be required to have experienced a pain intensity of at least 40mm on a 100-mm visual analogue scale in the most severely affected joint during the 24 hours prior to randomization.
5. Adequate liver and kidney function

   * Adequate liver function : SGOT, SGPT must be within 1.5 x normal limit
   * Adequate kidney function : Serum creatinine must be within 1.5 x normal limit
6. Subjects must be able to read, understand and follow the study instructions
7. Subjects must agree to informed consent spontaneously.

Exclusion Criteria:

1. Subjects who are not using adequate birth control.
2. Pregnant or breast-feeding.
3. Subjects requiring Knee surgery within 1 year of screening anticipating any need for a surgical procedure during the study.
4. Secondary OA patients
5. Similar OA patients(ex. rheumatic arthritis, bursitis etc)
6. Treatment with intra-articular injections of systemic corticosteroids or hyaluronic acid in the prior 3 months.
7. Use of drugs or psychotropic medicine(methadone maintenance program, codeine, tramadol hydrochloride)
8. Anemia or coagulant disorder
9. Use of anticoagulants or lithium
10. Use of misoprostol or H2-blocker(including anti ulcer medicine)
11. Presence or history of gastrointestinal bleeding within the past 1 year.
12. Subjects who have serious problem with cardiovascular, respiratory, endocrine, central nervous or History of neurotic mental.
13. Active malignancy of any type(ex. lymphoma, multiple myeloma etc)
14. Use of any medication that will affect pain perception during the study period; physical therapy, corticosteroids, NSAIDs, asprin, topical analgesics.
15. Use of glucosamine, chondroitin during the study period.
16. Change of concomitant dose/use within 4 weeks.
17. Known allergy or hypersensitivity to medicine.
18. Subjects received hormone replacement therapy.
19. Use of any other investigational drug within 1 month prior to screening.
20. Investigators determines that it is not appropriate.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
K-WOMAC | Visit 6(8 week), baseline
  The primary endpoint will be the change in the sum of the K-WOMAC OA index at Visit 6(8 weeks) vs. baseline(Visit 2, 0 week).

SECONDARY OUTCOMES:
knee pain intensity assessment | baseline, Visit 4(4 week), Visit 6(8 week)
  The change from baseline to each day(4 week and 8 week). Subjects assess knee pain intensity by using 100mm VAS at each time.
Global assessment(regarding to disease activity) | Visit 4(4 week), Visit 6(8 week)
  The change from Visit 4 to Visit 6 using 100mm VAS. Each patient and investigator assess by using 100mm VAS.
K-WOMAC each domain assessment | baseline, Visit 6(8 week)
  The change from Visit 6(8 weeks) vs. baseline(Visit 2, 0 week) in the K-WOMAC each domain score.
  * K-WOMAC 3 domains: pain domain, stiffness domain, physical function domain
ESR & hs-CRP | baseline, Visit 4(4 week), Visit 6(8 week)
  The change from baseline to each day(Visit 4, Visit 6) using laboratory test.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Jae Cho, MD, Study Chair — Kyunghee University Medical Center; Myung-Chul Lee, MD, Principal Investigator — Seoul National University Hospital; We-Yeon Won, MD, Principal Investigator — Ajou University Medical Center
Locations (3):
- South Korea (3):
  - KyungHee University medical center, Seoul, Hoegi-dong, Dongdaemun-gu
  - Ajou University Medical Center, Gyeonggi-do, Woncheon-dong Yeongtong-gu, Suwon
  - Seoul National University Hospital, Seoul, Yongon-dong, Chongno-gu